CLINICAL TRIAL: NCT01444794
Title: A National, Prospective Cohort to Document the Effectiveness of One BoNT-A Injection Cycle Based on Attainment of Individual Person-centred Goals in Adult Subjects Suffering From Lower Limb Spasticity Following Stroke
Brief Title: Adult Subjects Suffering From Lower Limb Spasticity Following Stroke
Acronym: VALGAS
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-92-52120-159
Record Dates: First submitted 2011-09-27; First posted 2011-10-03 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Spasticity
Keywords: Lower limb spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of the protocol is to assess the responder rate as defined by the achievement of the primary goal from the Goal Attainment Scale following one botulinum toxin type-A (BoNT-A) injection cycle in accordance with routine practices.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from lower limb spasticity following stroke
* With at least a 12-week interval between the last BoNT-A injection and inclusion
* Decision already been agreed to inject BoNT-A

Exclusion Criteria:

* Documented positive antigenicity to botulinum toxin
* Any neuromuscular junction indication
* Severe muscle atrophy in any muscle to be injected
* Any other indication that might interfere with rehabilitation or the evaluation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Responder rate as defined by the achievement of the primary goal from the Goal Attainment Scale (GAS). | Between 1 and 3 months from inclusion
  Assessed using the Goal Attainment Scale (GAS).

SECONDARY OUTCOMES:
Overall attainment of treatment goals | Between 1 and 3 months from inclusion
  Assessed using the GAS T-Score.
The use of standardized outcome measures and their results (e.g. muscle tone reduction, pain scores, functional tests). | Up to 5 months
Description of injection practices (BoNT-A: doses, volume, injection points, electromyography, electrostimulation and ecography). | Up to 5 months
Global assessment of benefits by both the investigator and the subject (or guardian). | Up to 5 months
  Assessed using a 5-point scale - much worse/worse/unchanged/better/much better

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (24):
- Spain (24):
  - Hospital Maritimo de Oza, A Coruña
  - Hospital de Cruces, Barakaldo
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital de Bellvitge, Barcelona
  - Hospital Mutua de Terrassa, Barcelona
  - Hospital Sant Pau, Barcelona
  - Hospital Vall Hebron, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - Hospital de Magdalena, Castellon
  - Hospital de Gorliz, Gorraiz
  - Hospital Dr. Negrín, Las Palmas de Gran Canaria
  - Hospital Insular, Las Palmas de Gran Canaria
  - Hospital De la Fundación Jimenez, Madrid
  - Hospital la Paz, Madrid
  - Hospital La Princesa, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Morales Meseguer, Murcia
  - Hospital Ntra. Sra. De La Candelaria, Santa Cruz de Tenerife
  - Hospital de Valdecilla, Santander
  - Hospital La Fe, Valencia
  - Hospital Valencia al Mar, Valencia
  - Hospital Povisa, Vigo
  - Hospital Xeral de Vigo, Vigo